CLINICAL TRIAL: NCT07389460
Title: Intravenous rhPro-UK Versus Placebo Before Endovascular Thrombectomy For Stroke Patient With Large Vessel Occlusion In The Extended Time Window: the Randomized, Placebo-controlled, Double-blind Trial (BRIDGE-PUK EXTEND )
Brief Title: Intravenous rhPro-UK Before Stroke Thrombectomy in the Extended Time Window (BRIDGE-PUK EXTEND)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Tasly Pharmaceutical Group Co., Ltd (Industry); Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJTU1AF2026LSYY-0065; BRIDGE-PUK EXTEND (Other Grant/Funding Number: Tasly Pharmaceutical Group Co., Ltd.)
Record Dates: First submitted 2026-01-27; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Large Vessel Occlusion Stroke; Recombinant Human Prourokinase; Extended Time Window; Intravenous Thrombolytic Therapy; Endovascular Treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhPro-UK group (Experimental): Patients in this group will be treated with intravenous rhPro-UK and endovascular thrombectomy
  Interventions: Drug: Intravenous rhPro-UK; Procedure: Endovascular thrombectomy
- Placebo group (Placebo Comparator): Patients in this group will be treated with intravenous placebo and endovascular thrombectomy
  Interventions: Drug: Intravenous placebo; Procedure: Endovascular thrombectomy

INTERVENTIONS:
Drug: Intravenous rhPro-UK — Patients will receive intravenous rhPro-UK
  Other Names: Intravenous PUK; Intravenous recombinant human prourokinase
  Arms: rhPro-UK group
Drug: Intravenous placebo — Patients will receive intravenous placebo
  Other Names: Intravenous placebo (a visually identical substance without pharmacological activity)
  Arms: Placebo group
Procedure: Endovascular thrombectomy — Patients will receive endovascular thrombectomy
  Other Names: Endovascular treatment; Mechanical thrombectomy

SUMMARY:
This randomized, double-blind, placebo-controlled phase III clinical trial aims to evaluate the efficacy and safety of intravenous recombinant human Prourokinase (rhPro-UK) in acute ischemic stroke patients with large vessel occlusion presenting 4.5-24 hours after last known well. The study will address two primary questions: 1) Whether rhPro-UK enhances pre-thrombectomy reperfusion rates and improves 90-day functional outcomes compared to placebo; 2) Whether rhPro-UK increases the risk of symptomatic intracranial hemorrhage and mortality.

Participants will be randomized to receive an intravenous bolus of rhPro-UK or matching placebo, with a total dose of 35mg (15mg administered as an intravenous push within 5 minutes, and the remaining 20mg continuously infused intravenously over 30 minutes). Key assessments include repeat neuroimaging (CT/CTA or MRI/MRA) at 24 hours post-treatment to evaluate reperfusion, NIH Stroke Scale score at day 5-7, and modified Rankin Scale score assessment at 90 days. Safety monitoring will focus on hemorrhagic transformation and mortality events throughout the study period.

DETAILED DESCRIPTION:
This multicenter, phase III trial employs a randomized, double-blind, placebo-controlled design to investigate the therapeutic window extension for rhPro-UK in large vessel occlusion stroke. Eligible participants are adults with large vessel occlusion confirmed by vascular imaging (CTA/MRA), and salvageable brain tissue demonstrated by perfusion imaging (CTP/MRP) mismatch. Exclusion criteria include contraindications to thrombolysis, and large core infarction (>70 mL on CTP).

Patients will be randomized 1:1 to receive either rhPro-UK or placebo, with a total dose of 35mg (15mg administered as an intravenous push within 5 minutes, followed by the remaining 20 mg continuously infused intravenously over 30 minutes) . All participants will undergo endovascular thrombectomy.

The primary outcome is functional independence (mRS 0-2) at 90 days. Secondary outcomes include substantial reperfusion at initial angiogram, first-pass reperfusion, final infarct volume on hour 36 CT, etc. Safety outcomes include symptomatic intracranial hemorrhage per Heidelberg Bleeding Classification criteria within 36 hours, and 90-day mortality.

Safety monitoring includes independent adjudication of hemorrhagic events and all-cause mortality. A sample size of 820 participants provides 80% power to detect a 10% absolute difference in functional independence (α=0.05).

The trial incorporates centralized blinded outcome assessment and intention-to-treat analysis, with data oversight by an independent clinical events committee and data safety monitoring board.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Acute ischemic stroke presenting within 4.5-24 hours of last known well;
3. No significant pre-stroke functional disability: for age <80 years, pre-stroke modified Rankin scale (mRS) ≤2; for age ≥80 years, prestroke mRS ≤1;
4. Baseline NIHSS score ≥6;
5. Imaging criteria of BOTH:

1. Occlusion on CTA/MRA in one of the following vessels: M1/M2 segment of middle cerebral artery, A1 segment of anterior cerebral artery, V4 segment of vertebral artery, basilar artery, or P1 segment of posterior cerebral artery. For A1, or P1 occlusions, vessel diameter must be ≥0.75 mm; 2. For anterior circulation occlusion: CTP/MRP demonstrating mismatch ratio ≥1.8, absolute mismatch volume ≥15 mL, and ischemic core volume <70 mL; OR have a mismatch between the presence of an abnormal signal on MRI diffusion-weighted imaging and no visible signal change on FLAIR. For posterior circulation occlusion: pc-ASPECTS score ≥6.

6. Plan to received endovascular thrombectomy; 7. The patient or their legal representative provides written informed consent.

Exclusion Criteria:

1. Intracranial hemorrhage confirmed by CT/MRI;
2. Onset accompanied by epileptic seizures, resulting in questionable stroke diagnosis and inability to obtain an accurate baseline NIHSS score;
3. Women who are pregnant or breastfeeding, or have a positive serum β-HCG test upon admission;
4. Already received intravenous thrombolytic after index stroke;
5. History of prior intracranial hemorrhage, including cerebral parenchymal hemorrhage, subarachnoid hemorrhage, and subdural/extradural hematoma;
6. Active bleeding or bleeding tendency, such as gastrointestinal bleeding, urinary tract bleeding, retinal hemorrhage, etc., or presence of coagulation dysfunction;
7. History of major recent surgery or trauma, such as intracranial or spinal surgery within the past 3 months, major surgery within the past 2 weeks, or severe head trauma within the past 3 weeks;
8. Baseline blood glucose <2.8 mmol/L or >22.2 mmol/L;
9. Received low molecular weight heparin within 24 hours, or oral anticoagulants with an International Normalized Ratio (INR) >1.7, or thrombin inhibitors within 48 hours, among others;
10. Arterial tortuosity or other vascular anomalies precluding endovascular access to target vessel;
11. Pre-existing neurological/psychiatric disorders interfering with neurological assessment;
12. Space-occupying intracranial tumors (except for small meningiomas);
13. Intracranial aneurysm or arteriovenous malformation;
14. Terminal illness with life expectancy <6 months;
15. Concurrent participation in other investigation clinical trials;
16. Presence of other conditions deemed by the investigator as unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients functionally independent (mRS score 0 to 2) at 90 days | 90 days post-randomization
  The modified Rankin Scale (mRS) is employed to assess patients' activities of daily living and the degree of disability. It grades patients' functional ability on a scale from 0 to 6, with a score of 0 indicating no symptoms and 6 representing death. An mRS score of 0-2 indicates functional independence.

SECONDARY OUTCOMES:
Distribution of mRS scores at 90 days | 90 days post-randomization
  The Modified Rankin Scale (mRS) is employed to assess patients' activities of daily living and the degree of disability. It grades patients' functional ability on a scale from 0 to 6, with a score of 0 indicating no symptoms and 6 representing death. The mRS score reflects the neurological functional status of stroke patients.
Shift in mRS score at 90 days | 90 days post-randomization
  The modified Rankin Scale (mRS) is employed to assess patients' activities of daily living and the degree of disability. It grades patients' functional ability on a scale from 0 to 6, with a score of 0 indicating no symptoms and 6 representing death. An mRS score shift reflects the improvement in the patient's neurological function.
Proportion of excellent functional outcome (mRS score 0 to 1) at 90 days | 90 days post-randomization
  The modified Rankin Scale (mRS) is employed to assess patients' activities of daily living and the degree of disability. It grades patients' functional ability on a scale from 0 to 6, with a score of 0 indicating no symptoms and 6 representing death. An mRS score of 0-1 indicates excellent functional outcome.
Score on the EQ-5D-5L scale at 90 days | 90 days post-randomization
  The EuroQoL 5-Dimension 5-Level (EQ-5D-5L) is a standardized health-related quality of life measurement instrument developed by the EuroQoL Group, primarily used to assess an individual's health status across multiple dimensions and their overall quality of life. The EQ-5D-5L describes an individual's health state based on five dimensions: Mobility, Self-care, Usual activities, Pain/Discomfort, and Anxiety/Depression. Scores range from 0, representing "the worst imaginable health," to 100, representing "the best imaginable health."
Change in NIHSS score from baseline to 5-7 days post-procedure or at discharge | 5-7 days post-procedure or at discharge
  The National Institutes of Health Stroke Scale (NIHSS) is a tool designed for the rapid assessment of neurological deficit severity. Each item is scored from 0 to 4 based on the patient's performance, with a total score ranging from 0 to 42. A higher score indicates a more severe neurological deficit.
NIHSS score at 5-7 days post-procedure or at discharge | 5-7 days post-procedure or at discharge
  The National Institutes of Health Stroke Scale (NIHSS) is a tool designed for the rapid assessment of neurological deficit severity. Each item is scored from 0 to 4 based on the patient's performance, with a total score ranging from 0 to 42. A higher score indicates a more severe neurological deficit.
Final infarct volume on hour 36 NCCT | 36 hours post-randomization
  Infarct volume quantified via NCCT , with manual correction by certified radiologists.
Substantial reperfusion (defined as an eTICI grade of 2b50, 2b67, 2c, or 3) at initial angiogram | within 5 minutes at initial angiogram
  The expanded Thrombolysis In Cerebral Infarction (eTICI) reperfusion grading system is a 7-point scale: 0 indicates no reperfusion noted; 1, reduction in thrombus without filling of distal arterial branches; 2a, reperfusion of <50% of the territory; 2b50, a reperfusion of 50-66% of the territory; 2b67, a reperfusion of 67-89% of the territory;2c, near-complete perfusion with distal slow flow or presence of small cortical emboli; and 3, complete reperfusion. Successful reperfusion at initial angiogram prior to thrombectomy was defined as an eTICI grade of 2b50, 2b67, 2c, or 3 on the first intracranial angiogram.
Successful reperfusion (defined as an eTICI grade of 2b, 2c, or 3) at end-of-procedure angiography | 15 minutes after initial angiogram
  The expanded Thrombolysis In Cerebral Infarction (eTICI) reperfusion grading system is a 7-point scale: 0 indicates no reperfusion noted; 1, reduction in thrombus without filling of distal arterial branches; 2a, reperfusion of <50% of the territory; 2b50, a reperfusion of 50-66% of the territory; 2b67, a reperfusion of 67-89% of the territory;2c, near-complete perfusion with distal slow flow or presence of small cortical emboli; and 3, complete reperfusion. This outcome will be evaluate at the end of procedure.
Modified first-pass reperfusion | Perioperative (After artery puncture, but the start of procedure)
  defined as Expanded Treatment in Cerebral Infarction 2b50, 2b67, 2c, or 3 after the first thrombectomy pass
Time from arterial puncture to successful recanalization or final angiography | Intraoperative
  The time (in minutes) from arterial puncture to successful recanalization or the final angiogram, reflecting the duration of the procedure.
Proportion of balloon angioplasty or stent placement during endovascular treatment | Intraoperative
  Endovascular treatment includes procedures such as thrombectomy, balloon angioplasty, and stent placement. This outcome specifically focuses on the proportion of patients undergoing balloon angioplasty or stent placement during endovascular therapy.
Proportion of patients planned for but ultimately not receiving endovascular treatment | Perioperative (After artery puncture, but the start of procedure)
  Patients planned for endovascular treatment may fail to undergo the procedure due to various reasons, including economic factors, disagreement among legal representatives, and changes in clinical condition, among others. This outcome focuses on the proportion of patients who were scheduled to receive but ultimately did not undergo endovascular treatment.
Symptomatic intracranial hemorrhage within 36 hours | within 36 hours after endovascular treatment
  evaluate intracranial hemorrhage (Heidelberg classification)
Proportion of patients with parenchymal hematoma at 36 hours post-procedure | within 36 hours after endovascular treatment
  European Cooperative Acute Stroke Study (ECASS) classification: Hemorrhagic infarction (HI) is divided into: HI1: Small petechial hemorrhages along the margins of the infarct. HI2: Confluent or multiple scattered petechial hemorrhages within the infarcted area. Parenchymal hematoma (PH) is divided into: PH1: Hematoma occupying ≤30% of the infarcted area, with mild mass effect. PH2: Hematoma occupying >30% of the infarcted area, with significant mass effect. This outcome will be evaluate the proportion of patients with PH2-type (parenchymal hematoma type 2) at 36 hours postoperatively.
Mortality within 90 days | 90 days post-randomization
  evaluate death rate of the two treatment groups
Procedural-related complications | within 90 days
  evaluate complications
Severe adverse events | within 90 days
  evaluate any adverse events

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Loudi Central Hospital, Loudi, Hunan
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Shihezi University, Shihezi, Xinjiang Uygur Autonomous Region
  - Xuanwu Hospital Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
study data without patient information
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Related papers published 6 months later, the IPD will be shared
Access Criteria: rabbit1110@163.com